CLINICAL TRIAL: NCT05753943
Title: CLINICAL TRIAL PHASE II, MULTICENTRIC, NATIONAL, DOUBLE-BLIND, PARALLEL, RANDOMIZED, AND PLACEBO-CONTROLLED FOR EVALUATION OF THE IMPROVEMENT OF SLEEP QUALITY IN PARTICIPANTS OF RESEARCH WITH INSOMNIA DISORDER
Status: No longer available | Type: Expanded Access
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernando Morgadinho Santos Coelho, PI, Federal University of São Paulo
Other Study IDs: 0001
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: insomnia; sleep initiation disorder; sleep maintenance disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: QUALI — Medication 1 pill at night
  Other Names: QUALI 50; QUALI 75

SUMMARY:
QUALI-001 code Phase II. Multicentric type. Test Product (QUALI-50) and (QUALI-75). Control Placebo capsule Primary goal Evaluate the improvement in sleep quality through the evaluation comparison of Pittsburgh Sleep Quality Index Scale scores obtained in visit 04 (final) compared to visit 02.

Evaluate the impact of treatments on improving sleep quality and total sleep time through actigraphic evaluation obtained through the average of the data observed in the last 07 days of treatment, compared to the average of the data observed in the 07 days of the basal period.

Outcome: A significant reduction in the score on the Scale is expected Pittsburgh Sleep Quality Index.

A significant increase in sleep efficiency is expected and a significant decrease in sleep latency time and the number of arousals evaluated through actigraphy.

Design Multicenter, randomized, placebo-controlled, parallel, with three treatments, in which each patient will receive treatment.

Arm 01: Control Treatment: Sleep Hygiene + Basic Medications + Placebo Arm 02: Treatment Test 1: Sleep hygiene + Basic drugs + (QUALI-50) capsule with the biphasic delivery system.

Arm 03: Treatment Test 2: Sleep Hygiene + Basic Medications+ (QUALI-75) capsule with the biphasic delivery system.

Population Research participants of both sexes, diagnosed with Moderate or severe insomnia disorder.

Control Treatment: Sleep Hygiene + Basic Medications + Placebo Treatment Test 1: Sleep hygiene + Basic drugs + (QUALI-50) capsule with the biphasic delivery system Treatment Test 2: Sleep Hygiene + Basic Medications+ (QUALI-75) capsule with the biphasic delivery system Reviews of efficiency Sleep quality scales, actigraphic measures, and sleep diary sleep. Reviews of security Clinical examination, monitoring of adverse events, electrocardiogram, and laboratory tests.

Criteria of Inclusion Agreement to participate in the study, documented through signature of the TCLE. Research participants diagnosed with Insomnia Disorder moderate or severe (≥ 10 points on the Pittsburgh scale). Stable research participant with outpatient treatment for Insomnia disorder for at least 60 days from visit 01 (initial). Age above 40 years. Research participants of both genders. Research participants were able to understand and provide their consent and complete the sleep diary and scales. Research participants with the ability to handle the actigraph properly. Women of childbearing age should accept the use of contraception during the study period. Men should accept the use of barrier contraceptives during the study period.

Criteria of Exclusion Research participants who are using drugs like benzodiazepines or other anxiolytics that may induce/alter sleep. Research participant having made previous use of Trazodone for less than 90 days from visit 01 (initial). Research participants having used MAOIs during a period of up to 30 days from visit 01 (initial). Research participants using barbiturates. Research participants using Linezolid for up to 30 days from visit 01 (initial). Research participants with a history of hypersensitivity to drugs. Research participants with a history of prolonged erection or priapism, abnormal orgasm, urinary incontinence, retention urinary tract, erectile dysfunction, retrograde ejaculation, clitorism, hematuria, and pollakiuria. Research Participants with a History of Beverage Addiction alcohol at the discretion of the investigator. Research participants with a history of clinical disease at the discretion of the investigator may confound the study results or are significant for the safety of the research participant. Pregnant or breastfeeding women. Research participants with a history of psychiatric illness serious or uncontrolled may influence the ability of the research participant to respond to the procedures of the study. Research participants with a significant history of hypotension. Research participants with a history of angle-closure glaucoma closed, photophobia, diplopia, xerophthalmia, and eye pain.

Research participants with a history of thyroid dysfunction significant or uncontrolled.

Taking the following CNS depressant drugs:

Carbamazepine, Buprenorphine/opioids, Inducing substrates or CYP3A4 inhibitors, Digoxin, phenytoin, Warfarin. Participants with prostatic hyperplasia.

Size of sample: Inclusion of approximately 99 research participants, divided into 3 parallel arms.

DETAILED DESCRIPTION:
QUALI-001 code Phase II. Multicentric type. Test Product (QUALI-50) and (QUALI-75). Control Placebo capsule Primary goal Evaluate the improvement in sleep quality through the evaluation comparison of Pittsburgh Sleep Quality Index Scale scores obtained in visit 04 (final) compared to visit 02.

Evaluate the impact of treatments on improving sleep quality and total sleep time through actigraphic evaluation obtained through the average of the data observed in the last 07 days of treatment, compared to the average of the data observed in the 07 days of the basal period.

Outcome: A significant reduction in the score on the Scale is expected Pittsburgh Sleep Quality Index.

A significant increase in sleep efficiency is expected and a significant decrease in sleep latency time and the number of arousals evaluated through actigraphy.

Design Multicenter, randomized, placebo-controlled, parallel, with three treatments, in which each patient will receive treatment.

Arm 01: Control Treatment: Sleep Hygiene + Basic Medications + Placebo Arm 02: Treatment Test 1: Sleep hygiene + Basic drugs + (QUALI-50) capsule with the biphasic delivery system.

Arm 03: Treatment Test 2: Sleep Hygiene + Basic Medications+ (QUALI-75) capsule with the biphasic delivery system.

Population Research participants of both sexes, diagnosed with Moderate or severe insomnia disorder.

Control Treatment: Sleep Hygiene + Basic Medications + Placebo Treatment Test 1: Sleep hygiene + Basic drugs + (QUALI-50) capsule with the biphasic delivery system Treatment Test 2: Sleep Hygiene + Basic Medications+ (QUALI-75) capsule with the biphasic delivery system Reviews of efficiency Sleep quality scales, actigraphic measures, and sleep diary sleep. Reviews of security Clinical examination, monitoring of adverse events, electrocardiogram, and laboratory tests.

Criteria of Inclusion Agreement to participate in the study, documented through signature of the TCLE. Research participants diagnosed with Insomnia Disorder moderate or severe (≥ 10 points on the Pittsburgh scale). Stable research participant with outpatient treatment for Insomnia disorder for at least 60 days from visit 01 (initial). Age above 40 years. Research participants of both genders. Research participants were able to understand and provide their consent and complete the sleep diary and scales. Research participants with the ability to handle the actigraph properly. Women of childbearing age should accept the use of contraception during the study period. Men should accept the use of barrier contraceptives during the study period.

Criteria of Exclusion Research participants who are using drugs like benzodiazepines or other anxiolytics that may induce/alter sleep. Research participant having made previous use of Trazodone for less than 90 days from visit 01 (initial). Research participants having used MAOIs during a period of up to 30 days from visit 01 (initial). Research participants using barbiturates. Research participants using Linezolid for up to 30 days from visit 01 (initial). Research participants with a history of hypersensitivity to drugs. Research participants with a history of prolonged erection or priapism, abnormal orgasm, urinary incontinence, retention urinary tract, erectile dysfunction, retrograde ejaculation, clitorism, hematuria, and pollakiuria. Research Participants with a History of Beverage Addiction alcohol at the discretion of the investigator. Research participants with a history of clinical disease at the discretion of the investigator may confound the study results or are significant for the safety of the research participant. Pregnant or breastfeeding women. Research participants with a history of psychiatric illness serious or uncontrolled may influence the ability of the research participant to respond to the procedures of the study. Research participants with a significant history of hypotension. Research participants with a history of angle-closure glaucoma closed, photophobia, diplopia, xerophthalmia, and eye pain.

Research participants with a history of thyroid dysfunction significant or uncontrolled.

Taking the following CNS depressant drugs:

Carbamazepine, Buprenorphine/opioids, Inducing substrates or CYP3A4 inhibitors, Digoxin, phenytoin, Warfarin. Participants with prostatic hyperplasia.

Size of sample: Inclusion of approximately 99 research participants, divided into 3 parallel arms.

ELIGIBILITY:
Inclusion Criteria:

Agreement to participate in the study, documented through the signature of the TCLE. Research participants diagnosed with Insomnia Disorder moderate or severe (≥ 10 points on the Pittsburgh scale). Stable research participant with outpatient treatment for Insomnia disorder for at least 60 days from visit 01 (initial). Age above 40 years. Research participants of both genders. Research participants were able to understand and provide their consent and complete the sleep diary and scales. Research participants with the ability to handle the actigraph properly. Women of childbearing age should accept the use of contraception during the study period. Men should accept the use of barrier contraceptives during the study period.

Exclusion Criteria:

Research participants who are using drugs like benzodiazepines or other anxiolytics that may induce/alter sleep. Research participant having made previous use of Trazodone for less than 90 days from visit 01 (initial). Research participants having used MAOIs during a period of up to 30 days from visit 01 (initial). Research participants using barbiturates. Research participants using Linezolid for up to 30 days from visit 01 (initial). Research participants with a history of hypersensitivity to drugs. Research participants with a history of prolonged erection or priapism, abnormal orgasm, urinary incontinence, retention urinary tract, erectile dysfunction, retrograde ejaculation, clitorism, hematuria, and pollakiuria. Research Participants with a History of Beverage Addiction alcohol at the discretion of the investigator. Research participants with a history of clinical disease at the discretion of the investigator may confound the study results or are significant for the safety of the research participant. Pregnant or breastfeeding women. Research participants with a history of psychiatric illness serious or uncontrolled may influence the ability of the research participant to respond to the procedures of the study. Research participants with a significant history of hypotension. Research participants with a history of angle-closure glaucoma closed, photophobia, diplopia, xerophthalmia, and eye pain.

Research participants with a history of thyroid dysfunction significant or uncontrolled. Taking the following CNS depressant drugs: Carbamazepine, Buprenorphine/opioids, Inducing substrates or CYP3A4 inhibitors, Digoxin, phenytoin, Warfarin. Participants with prostatic hyperplasia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Arriaga F, Cavaglia F, Pires AM, Lam E, Paiva T. Effects of trazodone on insomnia and anxiety in depressed patients: a clinical and sleep EEG study. Int J Psychiatry Clin Pract. 1997;1(4):281-6. doi: 10.3109/13651509709024740. PMID 24946195
- [Background] Ather SA, Ankier SI, Middleton RS. A double-blind evaluation of trazodone in the treatment of depression in the elderly. Br J Clin Pract. 1985 May;39(5):192-9. No abstract available. PMID 3907684
- [Background] Blacker R, Shanks NJ, Chapman N, Davey A. The drug treatment of depression in general practice: a comparison of nocte administration of trazodone with mianserin, dothiepin and amitriptyline. Psychopharmacology (Berl). 1988;95 Suppl:S18-24. doi: 10.1007/BF00172625. PMID 3133708
- [Background] Botros WA, Ankier SI, Priest RG, McManus IC, Steinert J, Samir ZY. Clinical assessment and performance tasks in depression: a comparison of amitriptyline and trazodone. Br J Psychiatry. 1989 Oct;155:479-82. doi: 10.1192/bjp.155.4.479. PMID 2692763
- [Background] Eraslan D, Ertekin E, Ertekin BA, Ozturk O. Treatment of insomnia with hypnotics resulting in improved sexual functioning in post-menopausal women. Psychiatr Danub. 2014 Dec;26(4):353-7. PMID 25377370
- [Background] Khazaie H, Ghadami MR, Knight DC, Emamian F, Tahmasian M. Insomnia treatment in the third trimester of pregnancy reduces postpartum depression symptoms: a randomized clinical trial. Psychiatry Res. 2013 Dec 30;210(3):901-5. doi: 10.1016/j.psychres.2013.08.017. Epub 2013 Aug 30. PMID 23993464